CLINICAL TRIAL: NCT06921603
Title: Point-of-Care Ultrasound-Guided Diuresis for Acute Decompensated Heart Failure to Reduce 30-Day Readmissions and Acute Kidney Injury
Brief Title: POCUS-Guided Diuresis for Decompensated Heart Failure
Acronym: POCUSHF-GD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, John Pacella, Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: STUDY24090092; 25POST1361664 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Heart Decompensation, Acute; Acute Kidney Injuries
Keywords: heart failure; point-of-care-ultrasound; readmission; acute kidney injury
MeSH Terms: conditions — Heart Failure; Acute Kidney Injury | interventions — Furosemide; Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two groups: a POCUS-assessed group and a standard care control group. Each group follows separate management protocols during the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- POCUS-assessed diuretic management (Experimental): Participants in this group will undergo daily POCUS imaging to assess volume status. The right internal jugular vein (RIJV) Distensibility Index (DI) will be measured and shared with the clinical team to guide diuretic (intravenous furosemide) management. However, all treatment decisions will be made at the discretion of the treating physicians.
  Interventions: Other: POCUS-Assessed Diuretic Management
- Furosemide (Standard Diuretic) Treatment (Active Comparator): Participants in this group will receive intravenous furosemide (standard diuretic) treatment, as part of their routine care, based on clinical evaluation. POCUS imaging will be performed daily for research only, and findings will not be shared with the clinical team. Treatment decisions will follow usual care protocols.
  Interventions: Other: Furosemide (Standard Diuretic) Treatment

INTERVENTIONS:
Other: Furosemide (Standard Diuretic) Treatment — Participants in this group will receive intravenous furosemide as part of their routine care, based on clinical assessments including symptoms, physical examination. Daily POCUS imaging will be performed for research purposes; however, the findings will not be shared with the treating clinical team. Fluid management decisions and discharge planning will follow usual care protocols, without additional imaging-based guidance.
  Arms: Furosemide (Standard Diuretic) Treatment
Other: POCUS-Assessed Diuretic Management — POCUS will be used to provide objective, non-invasive assessments of fluid status by measuring right internal jugular vein (RIJV) cross-sectional area (CSA) and calculating the Distensibility Index (DI). This information will be shared with the treating clinical team as an additional tool for fluid management. However, all final decisions regarding diuretic therapy will be made at the discretion of the treating physicians.
  Arms: POCUS-assessed diuretic management

SUMMARY:
Heart failure occurs when the heart cannot pump blood effectively, leading to fluid buildup in the body. This can cause problems such as difficulty breathing, swelling, and extreme tiredness. In severe cases, these symptoms worsen to the point where hospitalization is required. Unfortunately, many patients with severe heart failure are readmitted to the hospital within 30 days after discharge, which is both physically and emotionally challenging for patients and places a significant financial burden on individuals and the healthcare system.

Although symptoms such as difficulty breathing and swelling may improve during the hospital stay, some patients are discharged with excess fluid remaining in their bodies. This retained fluid often causes symptoms to worsen, leading to subsequent hospital readmissions. Inadequate management of fluid levels can also harm the kidneys, further complicating the patient's condition.

This study aims to improve care for heart failure patients by utilizing a simple, non-invasive tool to assess fluid levels more accurately at the bedside. The tool measures the size of a large blood vessel in the neck, providing key information about the pressure inside the heart. This information enables clinicians to determine the appropriate amount of medication needed to remove just the right amount of fluid. Properly managing fluid levels can help prevent kidney damage and improve overall patient outcomes.

The primary goal of this study is to evaluate whether this tool can reduce the number of patients readmitted to the hospital within 30 days of discharge. A secondary goal is to determine whether the tool can help protect kidney function by allowing for better fluid management. If successful, this approach has the potential to help heart failure patients stay healthier, reduce hospital visits, and lower healthcare costs.

DETAILED DESCRIPTION:
Heart failure is a major cause of hospitalization in the United States, affecting over 5 million adults, with 30-day readmission rates as high as 22%. Hospitalizations account for the majority of acute decompensated heart failure (ADHF)-related healthcare costs, and institutions that care for lower-income populations face added pressure under value-based payment models such as the Hospital Readmission Reduction Program (HRRP).

ADHF is characterized by elevated cardiac filling pressures and systemic congestion. Traditional clinical assessments, such as physical examination, chest radiography, and jugular venous pressure (JVP) evaluation, are often limited by low accuracy and high interobserver variability. Residual congestion at discharge is a key predictor of readmission and contributes to complications like acute kidney injury (AKI), which can occur in up to 20% of ADHF hospitalizations and is associated with increased mortality, longer length of stay, and higher healthcare costs (up to $80,400 per patient).

Point-of-care ultrasound (POCUS) has emerged as a valuable bedside tool for non-invasive, real-time volume assessment. This study focuses on a novel application of POCUS that uses the right internal jugular vein (RIJV) to estimate right atrial pressure (RAP). By measuring the cross-sectional area (CSA) of the RIJV during rest and the Valsalva maneuver, the Distensibility Index (DI) can be calculated. A DI ≥66% is associated with low RAP (≤12 mmHg), while lower values indicate persistent venous congestion.

Previous studies support the utility of this method. In a right heart catheterization cohort (n=67), DI predicted elevated RAP with 87% positive predictive value. In a prospective observational cohort (n=274), a DI ≥66% at discharge was associated with a 91.1% negative predictive value for avoiding early readmission. Patients with elevated RAP at discharge were 3.5 times more likely to be readmitted within 30 days.

This study introduces POCUS-guided diuretic management in hospitalized ADHF patients. The ultrasound-derived DI will be used to inform decisions regarding diuretic therapy and discharge readiness. All ultrasound operators will receive standardized training to ensure reproducibility of measurements. Clinician adherence to POCUS-guided recommendations will be monitored, and structured feedback will be obtained to assess usability.

By enhancing volume status assessment, this approach aims to improve decongestion strategies, reduce 30-day readmissions, and prevent kidney injury. If successful, this method could be integrated into routine clinical workflows, especially in settings where advanced imaging resources are limited. The study may inform future clinical guidelines and support more individualized, equitable care for patients with heart failure.

ELIGIBILITY:
List the inclusion criteria:

1. Age: Patients must be 18 years or older.
2. Diagnosis: Must have a confirmed diagnosis of acute decompensated heart failure (ADHF).
3. Treatment Plan: Patients must be planned for treatment with intravenous (IV) diuretics.
4. POCUS Measurement: Must have an abnormal right internal jugular vein (RIJV) distensibility index (DI) of <66% on point-of-care ultrasound (POCUS) at the time of admission.

These criteria ensure that participants are appropriately selected for the study and are likely to benefit from POCUS-guided diuretic management.

List the exclusion criteria:

1. Left Ventricular Assist Devices (LVAD): Patients with LVADs will be excluded due to their unique hemodynamics, which may interfere with study assessments.
2. Anatomical Incompatibilities: Excludes patients with RIJV or superior vena cava thrombus, congenital heart disease, or severe tricuspid regurgitation, as these conditions may impair accurate POCUS measurements.
3. Cardiomyopathy: Patients with hypertrophic or infiltrative cardiomyopathy will be excluded.
4. End-of-Life Care: Patients receiving hospice care or comfort measures only will not be included in the study.
5. Advanced Cancer: Patients with metastatic cancer will be excluded.
6. Severe Liver Dysfunction: Patients with a MELD-Na score greater than 20, indicating severe liver dysfunction, will be excluded.
7. End stage chronic kidney disease
8. Inability to Provide Consent: Patients who are unable to provide informed consent, due to cognitive impairment or other reasons, will not be eligible.
9. Inotropic Support: Patients requiring inotropic support at the time of enrollment will be excluded, as they represent a more severe heart failure profile that may not be suitable for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2025-06-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
30-Day Readmission Rate in Acute Decompensated Heart Failure (ADHF) Patients | From date of hospital discharge until date of first readmission for heart failure or 30 days post-discharge, whichever comes first.
  The percentage of participants readmitted to the hospital within 30 days of discharge for heart failure-related issues. The outcome compares the readmission rates between the POCUS-assessed diuretic management group and the standard care group.
Incidence of Acute Kidney Injury (AKI) | From baseline to hospital discharge and up to 30 days post-discharge (if readmitted).
  The percentage of participants who develop acute kidney injury (AKI) during hospitalization or within 30 days post-discharge (if readmitted).
  Definition: AKI will be defined using the Acute Kidney Injury Network (AKIN) criteria:
  * Increase in serum creatinine by ≥0.3 mg/dL within 48 hours OR
  * Increase in serum creatinine by ≥50% from baseline OR
  * Reduced urine output (<0.5 mL/kg/hr for ≥6 hours).
  Outcome Type: Binary (Yes/No)

SECONDARY OUTCOMES:
30-Day Mortality | From date of hospital discharge until date of death from any cause or 30 days post-discharge, whichever comes first.
  The percentage of participants who die within 30 days of discharge. This outcome compares mortality rates between the POCUS-assessed and standard care groups.
Length of Hospital Stay | From the date of hospital admission until the date of hospital discharge, assessed up to 60 days.
  The duration of hospitalization in days, measured for both groups.
Renal Function at Discharge | From date of hospital admission (baseline assessment) until date of hospital discharge, assessed up to 60 days.
  Change in eGFR (mL/min/1.73m²) from baseline to discharge to assess kidney function.
Adherence to POCUS-Based Recommendations | From date of hospital admission until date of hospital discharge, assessed up to 60 days.
  Percentage of cases in the POCUS-Assessed Group where clinicians followed POCUS-based recommendations for diuretic management.

CONTACTS AND LOCATIONS:
Overall Officials: John J Pacella, MD, Principal Investigator — University of Pittsburgh Medical Center (UPMC)
Locations (3):
- United States (3):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) collected in this study, including baseline characteristics, clinical outcomes, and POCUS measurements, will be shared. Data will be available upon reasonable request for researchers conducting methodologically sound studies that align with the objectives of this research.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and supporting documents will be available starting 6 months after publication of the primary results and will remain accessible for 5 years thereafter.
Access Criteria: Access to the dataset will be granted to researchers upon submission of a formal request, outlining the study objectives and analysis plan. Approval will be contingent upon compliance with ethical guidelines, data privacy regulations, and institutional review board (IRB) requirements. Researchers will be required to sign a data-sharing agreement (DSA) before receiving access.

REFERENCES:
- [Background] Kim WR, Biggins SW, Kremers WK, Wiesner RH, Kamath PS, Benson JT, Edwards E, Therneau TM. Hyponatremia and mortality among patients on the liver-transplant waiting list. N Engl J Med. 2008 Sep 4;359(10):1018-26. doi: 10.1056/NEJMoa0801209. PMID 18768945
- [Background] Abstract 12544: Point-of-Care Ultrasound Estimation of Right Atrial Pressure Predicts Early Readmission in Patients With Acute Decompensated Heart Failure
- [Background] Heldeweg MLA, Jagesar AR, Haaksma ME, Smit JM, Paulus F, Schultz MJ, Tuinman PR. Effects of Lung Ultrasonography-Guided Management on Cumulative Fluid Balance and Other Clinical Outcomes: A Systematic Review. Ultrasound Med Biol. 2021 May;47(5):1163-1171. doi: 10.1016/j.ultrasmedbio.2021.01.024. Epub 2021 Feb 23. PMID 33637390
- [Background] Yampolsky S, Kwan A, Cheng S, Kedan I. Point of Care Ultrasound for Diagnosis and Management in Heart Failure: A Targeted Literature Review. POCUS J. 2024 Apr 22;9(1):117-130. doi: 10.24908/pocus.v9i1.16795. eCollection 2024. PMID 38681155
- [Background] Chaudhary R, Sukhi A, Simon MA, Villanueva FS, Pacella JJ. Role of Internal Jugular Venous Ultrasound in suspected or confirmed Heart Failure: A Systematic Review. J Card Fail. 2022 Apr;28(4):639-649. doi: 10.1016/j.cardfail.2021.08.009. Epub 2021 Aug 19. PMID 34419599
- [Background] Allen LA, Smoyer Tomic KE, Smith DM, Wilson KL, Agodoa I. Rates and predictors of 30-day readmission among commercially insured and Medicaid-enrolled patients hospitalized with systolic heart failure. Circ Heart Fail. 2012 Nov;5(6):672-9. doi: 10.1161/CIRCHEARTFAILURE.112.967356. Epub 2012 Oct 16. PMID 23072736
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2022 May 3;79(17):e263-e421. doi: 10.1016/j.jacc.2021.12.012. Epub 2022 Apr 1. PMID 35379503
- [Background] Njoroge JN, Teerlink JR. Pathophysiology and Therapeutic Approaches to Acute Decompensated Heart Failure. Circ Res. 2021 May 14;128(10):1468-1486. doi: 10.1161/CIRCRESAHA.121.318186. Epub 2021 May 13. PMID 33983837
- [Background] Heidenreich PA, Fonarow GC, Opsha Y, Sandhu AT, Sweitzer NK, Warraich HJ; HFSA Scientific Statement Committee Members Chair. Economic Issues in Heart Failure in the United States. J Card Fail. 2022 Mar;28(3):453-466. doi: 10.1016/j.cardfail.2021.12.017. Epub 2022 Jan 24. PMID 35085762
- [Background] Psotka MA, Fonarow GC, Allen LA, Joynt Maddox KE, Fiuzat M, Heidenreich P, Hernandez AF, Konstam MA, Yancy CW, O'Connor CM. The Hospital Readmissions Reduction Program: Nationwide Perspectives and Recommendations: A JACC: Heart Failure Position Paper. JACC Heart Fail. 2020 Jan;8(1):1-11. doi: 10.1016/j.jchf.2019.07.012. Epub 2019 Oct 9. PMID 31606360
- [Background] Lahewala S, Arora S, Tripathi B, Panaich S, Kumar V, Patel N, Savani S, Dave M, Varma Y, Badheka A, Deshmukh A, Gidwani U, Gopalan R, Briasoulis A. Heart failure: Same-hospital vs. different-hospital readmission outcomes. Int J Cardiol. 2019 Mar 1;278:186-191. doi: 10.1016/j.ijcard.2018.12.043. Epub 2018 Dec 15. PMID 30579719
- [Background] Urbich M, Globe G, Pantiri K, Heisen M, Bennison C, Wirtz HS, Di Tanna GL. A Systematic Review of Medical Costs Associated with Heart Failure in the USA (2014-2020). Pharmacoeconomics. 2020 Nov;38(11):1219-1236. doi: 10.1007/s40273-020-00952-0. PMID 32812149
- [Background] Lala A, McNulty SE, Mentz RJ, Dunlay SM, Vader JM, AbouEzzeddine OF, DeVore AD, Khazanie P, Redfield MM, Goldsmith SR, Bart BA, Anstrom KJ, Felker GM, Hernandez AF, Stevenson LW. Relief and Recurrence of Congestion During and After Hospitalization for Acute Heart Failure: Insights From Diuretic Optimization Strategy Evaluation in Acute Decompensated Heart Failure (DOSE-AHF) and Cardiorenal Rescue Study in Acute Decompensated Heart Failure (CARESS-HF). Circ Heart Fail. 2015 Jul;8(4):741-8. doi: 10.1161/CIRCHEARTFAILURE.114.001957. Epub 2015 Jun 3. PMID 26041600
- [Background] Maw AM, Lucas BP, Sirovich BE, Soni NJ. Discharge-ready volume status in acute decompensated heart failure: a survey of hospitalists. J Community Hosp Intern Med Perspect. 2020 Jun 14;10(3):199-203. doi: 10.1080/20009666.2020.1759867. PMID 32850065
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Background] Metra M, Cotter G, Gheorghiade M, Dei Cas L, Voors AA. The role of the kidney in heart failure. Eur Heart J. 2012 Sep;33(17):2135-42. doi: 10.1093/eurheartj/ehs205. Epub 2012 Aug 10. PMID 22888113
- [Background] Mullens W, Abrahams Z, Francis GS, Sokos G, Taylor DO, Starling RC, Young JB, Tang WHW. Importance of venous congestion for worsening of renal function in advanced decompensated heart failure. J Am Coll Cardiol. 2009 Feb 17;53(7):589-596. doi: 10.1016/j.jacc.2008.05.068. PMID 19215833
- [Background] Romero-Gonzalez G, Manrique J, Slon-Roblero MF, Husain-Syed F, De la Espriella R, Ferrari F, Bover J, Ortiz A, Ronco C. PoCUS in nephrology: a new tool to improve our diagnostic skills. Clin Kidney J. 2022 Sep 12;16(2):218-229. doi: 10.1093/ckj/sfac203. eCollection 2023 Feb. PMID 36755847
- [Background] Simon MA, Kliner DE, Girod JP, Moguillansky D, Villanueva FS, Pacella JJ. Detection of elevated right atrial pressure using a simple bedside ultrasound measure. Am Heart J. 2010 Mar;159(3):421-7. doi: 10.1016/j.ahj.2010.01.004. PMID 20211304
- [Background] Simon MA, Schnatz RG, Romeo JD, Pacella JJ. Bedside Ultrasound Assessment of Jugular Venous Compliance as a Potential Point-of-Care Method to Predict Acute Decompensated Heart Failure 30-Day Readmission. J Am Heart Assoc. 2018 Aug 7;7(15):e008184. doi: 10.1161/JAHA.117.008184. PMID 30371245
- [Background] Doshi R, Dhawan T, Rendon C, Rodriguez MA, Al-Khafaji JF, Taha M, Win TT, Gullapalli N. Incidence and implications of acute kidney injury in patients hospitalized with acute decompensated heart failure. Intern Emerg Med. 2020 Apr;15(3):421-428. doi: 10.1007/s11739-019-02188-z. Epub 2019 Nov 4. PMID 31686359
- [Background] Cook DJ. Clinical assessment of central venous pressure in the critically ill. Am J Med Sci. 1990 Mar;299(3):175-8. doi: 10.1097/00000441-199003000-00006. PMID 2316561
- [Background] Gheorghiade M, Vaduganathan M, Fonarow GC, Bonow RO. Rehospitalization for heart failure: problems and perspectives. J Am Coll Cardiol. 2013 Jan 29;61(4):391-403. doi: 10.1016/j.jacc.2012.09.038. Epub 2012 Dec 5. PMID 23219302
- [Background] Lawson CA, Benson L, Squire I, Zaccardi F, Ali M, Hand S, Kadam U, Tay WT, Dahlstrom U, Lund LH, Savarese G, Lam CSP, Khunti K, Stromberg A. Changing health related quality of life and outcomes in heart failure by age, sex and subtype. EClinicalMedicine. 2023 Sep 14;64:102217. doi: 10.1016/j.eclinm.2023.102217. eCollection 2023 Oct. PMID 37745020
- [Background] Johansson I, Joseph P, Balasubramanian K, McMurray JJV, Lund LH, Ezekowitz JA, Kamath D, Alhabib K, Bayes-Genis A, Budaj A, Dans ALL, Dzudie A, Probstfield JL, Fox KAA, Karaye KM, Makubi A, Fukakusa B, Teo K, Temizhan A, Wittlinger T, Maggioni AP, Lanas F, Lopez-Jaramillo P, Silva-Cardoso J, Sliwa K, Dokainish H, Grinvalds A, McCready T, Yusuf S; G-CHF Investigators. Health-Related Quality of Life and Mortality in Heart Failure: The Global Congestive Heart Failure Study of 23 000 Patients From 40 Countries. Circulation. 2021 Jun;143(22):2129-2142. doi: 10.1161/CIRCULATIONAHA.120.050850. Epub 2021 Apr 28. PMID 33906372
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Heidenreich PA, Albert NM, Allen LA, Bluemke DA, Butler J, Fonarow GC, Ikonomidis JS, Khavjou O, Konstam MA, Maddox TM, Nichol G, Pham M, Pina IL, Trogdon JG; American Heart Association Advocacy Coordinating Committee; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Stroke Council. Forecasting the impact of heart failure in the United States: a policy statement from the American Heart Association. Circ Heart Fail. 2013 May;6(3):606-19. doi: 10.1161/HHF.0b013e318291329a. Epub 2013 Apr 24. PMID 23616602
- [Background] Patel J. Heart failure population health considerations. Am J Manag Care. 2021 Jun;27(9 Suppl):S191-S195. doi: 10.37765/ajmc.2021.88673. PMID 34042417